CLINICAL TRIAL: NCT02606058
Title: A Randomised Two Arm Open Label Controlled Trial Comparing Standard Immediate Cord Clamping Versus Deferring Cord Clamping for 60 Seconds or More in Babies Born Less Than 30 Weeks of Gestation to Determine Which Cord Clamping Method Results in Improved Survival and Less Disability.
Brief Title: The Australian Placental Transfusion Study (APTS): Should Very Pre Term Babies Receive a Placental Blood Transfusion at Birth Via Deferring Cord Clamping Versus Standard Cord Clamping Procedures?
Acronym: APTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-34236; ACTRN12610000633088 (Registry Identifier: Australian New Zealand Clinical Trials Registry)
Record Dates: First submitted 2015-01-08; First posted 2015-11-17 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early cord clamping (Control Arm) (No Intervention): Immediate cord clamping (< 10 seconds after birth). The cord is clamped 6 cm from the umbilicus within ten seconds of delivery of the baby.
- Deferred cord clamping (Experimental): Deferred cord clamping. Investigator/Research personnel holds the baby as low as possible below the level of the introitus or placenta for 60 seconds and not to exceed 80 seconds, then clamps the cord about 6 cm from the umbilicus.
  Interventions: Procedure: Deferred cord clamping

INTERVENTIONS:
Procedure: Deferred cord clamping — Deferred cord clamping (for 60 seconds or more with the baby held below or at the level of the placenta)
  Arms: Deferred cord clamping

SUMMARY:
To establish if placental transfusion, using deferred cord clamping for 60 seconds or more while holding the baby at or below the level of the placenta, will improve survival without disability compared with standard early cord clamping in preterm babies less than 30 weeks of gestation.

DETAILED DESCRIPTION:
Most preterm babies have the umbilical cord clamped within 10 seconds of birth. Placental transfusion is a simple way of giving the baby extra blood at birth by delaying the clamping of the umbilical cord by 60 seconds or more. There is promising evidence from randomised trials that placental transfusion in babies less than 37 weeks of pregnancy may improve their blood pressure, reduce the number of blood transfusions needed and decrease bleeding into the brain, bowel disease and infection. However, we not know if babies born before 30 weeks of pregnancy benefit or if placental transfusion increases or decreases death or childhood disability. Despite this uncertainty more doctors are recommending that all very preterm babies are given a placental transfusion at birth. It is important to find out if placental transfusion does more good than harm, before it becomes even more widely used.

The Australian Placental Transfusion Study will enrol at least 1600 women who will give birth to babies born less than 30 weeks of gestation. These participants will be randomly assigned to either standard treatment where the umbilical cord is clamped within 10 seconds of birth or a second method where the umbilical cord will be clamped after waiting for 60 seconds or more at birth while the baby is being held below the level of the placenta. The main research question is whether placental transfusion reduces death and disability when the baby is discharged from hospital and into childhood.

ELIGIBILITY:
Inclusion Criteria:

Women who have a reasonable chance of delivering less than 30 weeks of gestation. Informed consent has been received from the parent or guardian.

Exclusion Criteria:

No indication or contraindication to placental transfusion, in the view of mother or baby.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1637 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Death and/or major morbidity at 36 weeks post menstrual age | 36 weeks post menstrual age
  Composite death and/or major morbidity at 36 completed weeks post menstrual age. Morbidity is defined by one or more of the following: brain injury on ultrasound, severe retinopathy, necrotising enterocolitis, late onset sepsis.

SECONDARY OUTCOMES:
Incidence of death | 36 completed weeks post menstrual age
  The death component of the composite primary outcome
Incidence of major morbidity | 36 completed weeks post menstrual age
  Major morbidity (incidence of one or more of brain injury on ultrasound, severe retinopathy, necrotising enterocolitis or late onset sepsis).
Incidence of death or major disability | Up to 3 years corrected age
  Death or major disability (for example cerebral palsy with inability to walk; blindness; deafness; major problems with language or speech; ASQ score indicative of developmental delay)
Incidence of death or brain injury on ultrasound | 36 completed weeks post menstrual age
  Death or brain injury on ultrasound
Major disability defined as cerebral palsy with an inability to walk unassisted, severe visual loss, deafness, major problems with language or speech, or a score indicative of developmental delay on Ages and Stages Questionnaire. | Up to 3 years corrected age
Brain injury on ultrasound | 36 completed weeks post menstrual age
IVH (all grades) seen on ultrasound | 36 completed weeks post menstrual age
IVH (Grades 3 & 4) seen on ultrasound | 36 completed weeks post menstrual age
IVH (Grade 4) seen on ultrasound | 36 completed weeks post menstrual age
Severe retinopathy warranting treatment or Stage 4 retinopathy according to the Australian and New Zealand Neonatal Network (ANZNN) definitions | 36 completed weeks post menstrual age
Necrotizing enterocolitis with the following signs: at least 1 systemic sign, profile consistent with definite NEC, warranted treatment for NEC. | 36 completed weeks post menstrual age
Patent ductus arteriosis requiring treatment (documented in medical records) | 36 completed weeks post menstrual age
Chronic lung disease, defined as receiving supplemental oxygen or any form of assisted ventilation at 36 completed weeks post menstrual age for 4 consecutive hours in a 24 hour period | 36 completed weeks post menstrual age
Late onset sepsis, defined as a clinical picture consistent with sepsis, and either a positive culture of blood and/or CSF, or a positive urine culture by sterile collection, and at least 5 days of antibiotic treatment. | 36 completed weeks post menstrual age
Death up to 3 years corrected age | Up to 3 years corrected age

CONTACTS AND LOCATIONS:
Overall Officials: William T Mordi, MD, Principal Investigator — University of Sydney
Locations (26):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - University of Vermont Medical Centre, Burlington, Vermont
- Australia (14):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - John Hunter Hospital, Newcastle, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Royal Hospital for Women, Sydney, New South Wales
  - Nepean Hospital, Sydney, New South Wales
  - Mater Mother's Hospital, Brisbane, Queensland
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Townsville Hospital, Townsville, Queensland
  - Flinders Medical Centre, Adelaide, South Australia
  - Monash Medical Centre, Melbourne, Victoria
  - Mercy Hospital for Women, Melbourne, Victoria
  - King Edward Memorial Hospital, Perth, Western Australia
- IWK Health Center, Halifax, Nova Scotia, Canada
- Hôpital Antoine-Béclère, Clamart, France
- New Zealand (5):
  - Auckland Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton
  - Wellington Hospital, Wellington
- Aga Khan University Hospital, Karachi, Pakistan
- United Kingdom (2):
  - Royal Jubilee Maternity Hospital, Belfast, Northern Ireland
  - Craigavon Area Hospital, Craigavon, Northern Ireland